CLINICAL TRIAL: NCT02113722
Title: Does Left Cardiac Sympathectomy Stellate Ganglionectomy Confer an Added Benefit Over Optimal Medical Therapy in the Reduction of Therapy Delivered From an Implanted Cardioverter Defibrillator in Patients at High Risk of Sudden Cardiac Death
Brief Title: Is Left Stellate Ganglionectomy Beneficial to Patients With Life Threatening Ventricular Arrhythmias
Acronym: Reduce-SCD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study already undertaken at another centre
Sponsor: Cindy Hall (Other)
Responsible Party: Sponsor-Investigator, Cindy Hall, Dr Gerald Kaye, Princess Alexandra Hospital, Brisbane, Australia
Organization: Princess Alexandra Hospital, Brisbane, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14_145; Version 1 dated 12 March 2014 (Other: Princess Alexandra Hospital)
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Sudden Cardiac Death
Keywords: Sudden cardiac death; Ganglionectomy; Ventricular arrhythmia; Cardiac surgery; Implanted cardiac defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left cardiac sympathetic denervation (Active Comparator): Left cardiac sympathetic denervation
  Interventions: Procedure: Left cardiac sympathetic denervation
- Standard of care (Placebo Comparator): Continuing medical therapy
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Left cardiac sympathetic denervation — Left cardiac sympathetic denervation via a video
  Arms: Left cardiac sympathetic denervation
Procedure: Standard of Care — Medical therapy
  Arms: Standard of care

SUMMARY:
The purpose of this study is to determine whether the incidence of recurrent life threatening ventricular arrhythmias in patients with an implanted cardiac defibrillator (ICD) can be reduced if a surgical left stellate ganglionectomy is performed.

DETAILED DESCRIPTION:
Background: Sudden cardiac death (SCD) is a devastating problem. There is a strong body of evidence which suggests an important role of the autonomic nervous system in the genesis of sudden cardiac death. An increase in vagal tone improves cardiac electrical stability whereas sympathetic hyper-stimulation may precipitate ventricular fibrillation, particularly in the ischaemic heart.

In patients with life threatening ventricular arrhythmias an implanted cardiac defibrillator (ICD) is the treatment of choice. Ventricular arrhythmias can be terminated by either an intra-cardiac shock, often a painful therapy particularly if the patient should remain conscious, or by anti-tachycardia pacing (ATP) which is painless and often is unnoticed.

Despite intensive pharmacological treatment with beta-blockers and often amiodarone, patients may still have up to 20% risk per year of receiving an internal shock for both life threatening and sometimes for a non life threatening arrhythmia. A technique that might reduce the risk of shock delivery over and above current approaches would be an advantage.

It has been suggested that a surgical left stellate ganglionectomy (also referred to as left cardiac sympathetic denervation - LCSD) in patients cardiac arrhythmias may have potential antiarrhythmic benefit particularly in patients with life threatening ventricular arrhythmias and/or at high risk of sudden death (SCD) despite current medical therapy. Recent improvements in surgical techniques has allowed a video assisted minimal access approach (VATS) with a reduction in inpatient stay and increased patient tolerability. The overall risk profile is the same as open thoracotomy but at a much reduced rate.

Current data suggests that LCSD is a reasonable management option in patients with recurrent ventricular arrhythmias.

Hypothesis: Does VATS assisted LCSD in patients with an ICD implanted for secondary prevention, on chronic amiodarone therapy reduce shock frequency and anti-tachycardia pacing compared to optimal medical treatment - a prospective study.

Protocol: All patients with an ICD who present with an intra-cardiac shock or ATP for the termination of a ventricular arrhythmia (VT or VF) will be eligible for this study. All patients will be established on optimal medical treatment (angiotensin-converting-enzyme (ACE) inhibitor/angiotensin receptor blockers (ARB) and beta blockers) and amiodarone (unless documentation exists of amiodarone intolerance), for three months, as defined in inclusion criteria. Patients will be given the Participant Information Sheet describing the study and signed Informed Consent will be obtained.

Baseline tests will be performed in both groups. Patients will be randomised in a 1:1 fashion to either continued medical treatment or continued medical treatment plus minimal access video assisted left stellate ganglionectomy.

Surgery will be performed within two weeks of randomisation. Surgical patients will be discharged from hospital at the discretion of their treating surgeon. The surgical patients will be assessed in a clinic two weeks after discharge.

All patients will be followed for a total of 365 days from randomisation.

Primary Endpoint:

• Intra-cardiac shock frequency and frequency of anti-tachycardia pacing over a 12 month period commencing from time of randomisation to a minimum of 365 days post-study entry.

Secondary Endpoints:

* All-cause mortality
* Heart Failure hospital admissions after randomisation
* Early and late surgical complications -

  * death
  * Horner's syndrome
  * length of hospital stay
  * post-operative pain
  * sweating in the left hand and axilla
  * damage to brachial plexus
* Changes in heart rate variability (HRV)
* Inappropriate intra-cardiac shocks for atrial tachyarrhythmias: atrial fibrillation, flutter and tachycardia
* Changes in left ventricular function (ejection fraction) measured by echocardiography
* Changes in heart-to-mediastinum (H/M) ratio on iodine-131-meta-iodobenzineguanidine (MIBG)
* Alterations in the surface twelve lead ECG including:

  * change in the QT interval
  * changes in QT dispersion on the surface ECG
  * changes in QRS duration
  * Changes in ICD device derived parameters:
  * Frequency of non-sustained ventricular tachycardia and of ventricular premature contractions
  * Changes in heart rate variability
  * If appropriate (ICD dependent) changes in transthoracic impedance
  * Atrial fibrillation burden
  * Quality of life assessment (SF36)

Sample Size Sample size will be based upon a projected 10% shock rate in the first 12 months and a mortality of 5-8% (1,2,3). As this is a pilot study the sample will be 25 patients in each group (medical treatment alone vs. LCSD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18yrs old or older.
* Medical indication for an ICD for secondary prevention as per standard ESC/ACC guidelines.
* Patients with single, dual chamber or biventricular defibrillators (CRT-D) will be included.
* Intra-cardiac shock or ATP for VT or VF:

  * For study inclusion the patient must have had a recent intra-cardiac shock or ATP (≤30 days).
  * For study inclusion the patient must be on optimised amiodarone therapy (≥3 months) or have documented evidence of amiodarone intolerance.
  * For study inclusion the Intra-cardiac shock or ATP for VT or VF must not be secondary to a reversible biochemical or drug induced arrhythmia.
* Ejection fraction of ≤ 40% measured ≤ 6 months prior to the Baseline Visit.
* Surgical review to ensure patient is suitable for surgery.
* Women of childbearing potential must have a negative pregnancy test.
* Written informed consent.

Exclusion Criteria:

* Age less than 18years.
* Pregnancy.
* Predicted life expectancy of less than one year.
* Intra-cardiac shock or ATP for VT or VF secondary to a reversible biochemical or drug induced arrhythmia.
* Severe renal impairment with an estimated glomerular filtration rate (eGFR) of less than 20mL/mins.
* Unsuitable for cardiac surgery.
* Non-optimised heart failure medications (ACE inhibitors/ARB blockers and/or beta-blockers).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite outcome measure of intra-cardiac shock frequency and frequency of anti-tachycardia pacing | 12 months
  Hypothesis Does video assisted minimal access approach for left cardiac sympathetic denervation in patients with an ICD implanted and on amiodarone for secondary prevention at high risk of sudden death reduce shock frequency and anti-tachycardia pacing compared to optimal medical treatment - a prospective study.
  Primary End Point Intra-cardiac shock frequency and frequency of anti-tachycardia pacing over a 12 month period commencing from time of randomisation to a minimum of 365 days post-study entry.
  The ICD will be interrogated as per clinical practice prior to signing the Informed Consent form as well as at the 6 and 12 month study follow-up visits. The device will be interrogated within 24 hours of delivery of an intra-cardiac shock or if the patient feels there has been therapy delivery (e.g. ATP).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Kaye, MBBS, Study Chair — Princess Alexandra Hospital
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
Data is de-identified and will not be shared.